CLINICAL TRIAL: NCT03702114
Title: Detecting Auricular Points Among Patients With Menstrual Migraine by A Novel Auricular Point Detector (APD): A Pilot Diagnostic Accuracy Study
Brief Title: Detecting Auricular Points in MMG by a Novel APD ( APD-MMG )
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other); City University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: SCM-ACU-03
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Menstrual Migraine
Keywords: menstrual migraine; auricular point; diagnostic accuracy; Auricular Point Detection device

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MMG group: Patients in this group will receive auricular point detection which is accomplished by the novel auricular point detector device. There is no addition to the patient's routine care.
  Interventions: Device: auricular point detection
- Control group: This group includes healthy subject, for whom no treatment will be performed. Only auricular point detection by the auricular point detector will be conducted.
  Interventions: Device: auricular point detection

INTERVENTIONS:
Device: auricular point detection — This device is only for auricular detection. No additional intervention will be delivered.

SUMMARY:
This pilot study is designed to validate the diagnostic ability of a novel APD for auricular point detection among patients with menstrual migraine (MMG), as compared with an already commercialized device.

DETAILED DESCRIPTION:
This pilot study is designed to evaluate the diagnostic ability of a novel APD for auricular point detection among patients with menstrual migraine (MMG), as compared with an already commercialized device. The investigators will test if the novel APD could provide a more reliable and quantifiable diagnosis of MMG-related auricular point than traditional devices currently available in the market; The study will also use the APD device to test whether the cutaneous electrical impedance detected from the corresponding auricular points by the novel device is the lowest in the reproductive organ and facial area in the MMG population. As a pilot study, 12 patients with MMG will be recruited from the School of Chinese Medicine, the University of Hong Kong. 12 healthy subjects will be recruited from the university community. Auricular acupoint detection will be accomplished with the new device and a control device. The electrical impedance will be measured and recorded. Patient's condition will also be evaluated by the visual analogue scale (VAS) and the Modified New England Center of Headache (NECH) headache calendar. The specificity and sensitivity of the auricular point detection by the APD device will be calculated. Cohen's kappa coefficient (κ) will be used to test the inter-methods reliability, test-retest reliability, and inter-tester reliability. Moreover, the Pearson Correlation Coefficient will be used to test the correlation between the electrical impedance of the auricular point and the pain intensity score.

ELIGIBILITY:
Inclusion Criteria:

* When attacks, average migraine pain severity >=5 point measured by a 10-point VAS scale;
* Diagnosed pure menstrual migraine without aura or menstrually related migraine without aura according to The International Classification of Headache Disorders: 2nd edition;
* Provide written inform consent;
* Free of any other diagnosed psychological conditions;

Exclusion Criteria:

* with any other diseases such as cardiovascular, renal, neurological, digestive, hepatic, respiratory disease
* Pregnancy or lactation
* Participation in a clinical study that may interfere with participation in this study
* History of or current tobacco, alcohol use
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study
* Unable to provide written informed consent due to any reason.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only female subject will be included in this study because the disease investigated is menstrual migraine.
Study Population: Eligible menstrual migraine patients will be recruited from the Sassoon Road Clinic of the School of Chinese Medicine, the University of Hong Kong.
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2018-10-15 (Estimated); Primary Completion 2019-01-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
cohen's kappa coefficient | baseline
  The Cohen's kappa coefficient is a statistical test used to validate the inter-method reliability, test-retest reliability and inter-observer reliability of the device.

SECONDARY OUTCOMES:
the Visual Analogue Scale (VAS) | baseline
  The VAS is a common instrument used to measure pain intensity. The scale ranges from 0 to 10, where 0 indicates no pain and 10 indicates worst pain possible.
the Modified New England Center of Headache (NECH) headache calendar | baseline
  The Modified New England Center of Headache (NECH) headache calendar is a pain diary that can be used to record the time, frequency, intensity and relief of migraine attacks in a month. It employs a 0-10 numeric rating scale (NRS) to quantify the pain intensity of migraine. The frequency and the average pain intensity of menstrual migraine is calculated.
self-developed questionnaire on patient's attitude towards complementary therapies for pain management | baseline
  This is a self-developed questionnaire which includes 10 items aiming to survey patient's attitude towards the use of complementary therapies for pain management. This questionnaire only includes descriptive answers to be choose. The percentage for each choice will calculated.
The diagnostic specificity of the device | baseline
  The specificity test is a test to validate the ability of a diagnosis to tell the 'non-disease' among those without the disease.
The diagnostic sensitivity of the device | baseline
  The sensitivity test is a test to validate the ability of a diagnosis to tell the 'disease' among those with the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Lixing Lao, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, HKU, Hong Kong, INTL, Hong Kong

IPD SHARING:
Plan to Share IPD: No
IPD sharing will be at the discretion of the study-involved participants and the principal investigator.